CLINICAL TRIAL: NCT05263297
Title: The Effect of Two Different Cognitive-Behavioral Combined Programs in Blood Collection on Children's Pain, Fear and Anxiety and Parents' Satisfaction Level: A Randomized Controlled Study
Brief Title: The Effect of Two Different Cognitive-Behavioral Combined Programs in Blood Collection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Ayse Sonay Turkmen, Prof.Dr, Assoc.Prof., Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Cognitive-Behavioral
Record Dates: First submitted 2022-02-10; First posted 2022-03-02 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Child Behavior; Pain, Acute; Fear
MeSH Terms: conditions — Child Behavior; Acute Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video group (Other): During the bloodletting process, children in the video game group will be played with audio and visual video games that they can play with one hand. Thus, children will be provided with both visual and auditory stimuli. It will be preferred that children play the video game that they have knowledge about and know how to play the game. For this reason, children in the video game group will be given the chance to choose video games suitable for their age and development level on their parents' smartphones. These video games within the scope of the research will not be named and will not be promoted/advertised.
  Interventions: Other: control group
- kaleidoscope group (Other): In this study, a kaleidoscope with colorful patterns that can be used by children with one hand will be used. In the research, the kaleidoscope will be introduced to children and how to use it will be explained. After the procedure, the kaleidoscope will be disinfected using appropriate disinfectant materials.
  Interventions: Other: control group

INTERVENTIONS:
Other: control group — no intervention will be made.

SUMMARY:
The aim of this study is to investigate the effect of two different cognitive-behavioral combined programs, including video games or kaleidoscope, on the pain, fear and anxiety experienced by children who apply for therapeutic or diagnostic venous blood collection, and their parents' satisfaction levels. In addition, this research aims to create a holistic approach to child health due to the evaluation of both children and parents.

The population of the research will be children aged 8-10 who come to the Children's Blood Collection Unit of Karaman Training and Research Hospital between February 2022 and March 2022. The sample of the study will consist of 96 children and their parents who applied to the Blood Collection Unit on the specified dates, met the inclusion criteria and agreed to participate in the study. The pediatric blood collection unit provides service between 08:00 and 16:00 on weekdays. In order to determine the number of samples, power analysis was performed using the G*Power (v3.1.9) program. It was planned to carry out the research with a total of 96 children and their parents, 32 in each group, considering possible case losses during the research period.

Evaluation of the data will be done in the computer environment with the SPSS (Statistical Package for Social Sciences) 22.0 package program. Percentage distributions, mean, standard deviation, chi-square test, analysis of variance will be used in the analysis of the data. In addition, the variance of the groups will be examined with the Levene test in order to make further analysis. In cases where the variance is equal, Bonferroni analysis will be used in post hoc advanced analyses, and Dunnett T3 analysis will be used in cases where the variance is not equal. The research findings will be evaluated at the 95% confidence interval, at the p<0.05 significance level.

DETAILED DESCRIPTION:
Type of Research The study was planned in a randomized controlled experimental research design to examine the effect of two different cognitive-behavioral combined programs, including video games or kaleidoscope, on the pain, fear and anxiety experienced by children due to venous blood collection and the satisfaction levels of their parents.

Variables of the Study Dependent variables: Children's Visual Analog Scale (VAS), Wong Baker Faces Pain Scale (Wong-Baker Faces Pain Scale- W-BFS), Child Fear Inventory (CDS), Child Anxiety Scale-State Scale (CAS-D), PedsQL Health Scores from the Care Parental Satisfaction Scale.

Independent variables: Sociodemographic characteristics, video game or kaleidoscope, including two different cognitive-behavioral combined program applications.

Hypotheses Hypothesis 1. Cognitive-behavioral combined program including video game in blood collection has an effect on children's pain, fear and anxiety levels.

Hypothesis 2. Cognitive-behavioral combined program including kaleidoscope in blood collection has an effect on children's pain, fear and anxiety levels.

Hypothesis 3. There is a difference in pain, fear and anxiety levels between the children who used the cognitive-behavioral combined program including video game in blood collection and the children who used the cognitive-behavioral combined program including kaleidoscope.

Hypothesis 4. Cognitive-behavioral combined program including video game in blood collection has an effect on parents' satisfaction levels.

Hypothesis 5. Cognitive-behavioral combined program including kaleidoscope in blood collection has an effect on parents' satisfaction levels.

Hypothesis 6. There is a difference in satisfaction levels between the parents of the children who used the cognitive-behavioral combined program including video game in the blood collection process and the parents of the children who used the cognitive-behavioral combined program including the kaleidoscope.

In order to determine the number of samples, power analysis was performed using the G*Power (v3.1.9) program. The power of the study is expressed as 1-β (β = probability of type II error), and in general studies should have 80% power. Power analysis was performed to determine the adequacy of the sample size of the study; The power of the study was determined to be 0.95 with a significance level of 0.05, a confidence interval of 0.95, and an effect size of 0.97. Accordingly, there must be 29 people in each group. It was planned to carry out the research with a total of 96 children and their parents, 32 in each group, considering possible case losses during the research period.

Randomization The process of enrolling children and parents into groups will be randomly assigned. In the study, "stratification and block randomization methods" will be used in assigning participants to control and intervention groups. It has been reported in the literature that age, gender, and fear of interventional procedures are among the factors affecting the fear and stress experienced by children in interventional procedures. Accordingly, the children will be stratified as "girl and boy" for the gender variable, "afraid and not afraid" for the fear of the procedure, and randomization with blocks will be applied. The determined layers were created as codes obtained from the permutation-based computer program. At the beginning of the research, which letter would be the intervention or control group was determined by the closed opaque envelope method. Accordingly, the A was used for the control group, the B for the cognitive-behavioral combined program with the video game, and the C for the cognitive-behavioral combined program with the kaleidoscope. These block sets will be placed in envelopes of different colors and sizes by the researcher and kept in a black bag. It will be determined which stratum the children are in. It will be determined which group the determined child will be in according to the block set randomly drawn by the children from the black bag. The groups chosen by the children will be the same as those of their parents. If the next children are in the same layer, the block set will continue until the completion of the set. When it is determined that the incoming child is in a different layer, a new block set will be selected from the bag and the group will be determined.

S1 Girl, Afraid ABAA, CACB, ACBB, CABC, BACC, BACB S2 Girl, Not afraid AACB, ABAC, ABAB, CACB, BCCC, ABBC S3 Boy, Afraid ABCC, ABCA, BCAC, ABBB, CBBC, CAAA S4 Boy, Not afraid ABAA, CACB, ACBB, CABC, BCAB, ACCB

Venous blood collection of all children included in the study will be performed by an experienced nurse in the pediatric blood collection unit. Thus, the application differences that may occur during the venous blood collection process will be eliminated. It was planned to collect the information about the children and their families in a time period of approximately 5 minutes before the procedure by face-to-face interview method by the researcher using the "Descriptive Information Form". In addition, the researcher will introduce the measurement tools that they will score to children and parents.

According to the routine application of the blood collection unit, the features related to the blood collection process are listed below:

* The area where the venous blood sample is taken (thick in the antecubital fossa/ vein near the skin surface)
* The thickness of the needle used in the process (21 G 38 mm needle)
* Blood collection technique used (using the same type of tourniquet)
* Environmental factors (Heat, light and noise control)
* phlebotomy chair for children
* The antiseptic solution used (70% alcohol)
* Processing time (Average 3 minutes)

In data collection, Child and Parent Diagnosis Form, Children's Visual Analog Scale (VAS), Wong Baker Faces Pain Scale (Wong-Baker Faces Pain Scale- W-BFS), Child Fear Scale (CDS), Child Anxiety Scale-State Scale (CAS) were used. -D), two different cognitive-behavioral combined program applications including PedsQL Health Care Parental Satisfaction Scale, Video game or kaleidoscope will be used.

Child and Parent Identification Form The sample is a form prepared by the researcher by taking expert opinion and reviewing the literature to obtain information about the selected children and their parents. Form; it consists of questions that include the demographic characteristics of the child and his parents, whether the child has any disease, and the variables that may affect the child's pain and fear levels due to the procedure. Before starting the research, the interview and observation form will be applied to five children and their parents. Incomprehensible parts will be corrected and finalized. These children and their parents will be excluded from the research.

Visual Analog Scale (VAS-Visual Analog Scale) The VAS is usually presented as a 10 cm line with one end marked 'no pain' and the other 'worst imaginable pain'. Patients are asked to mark the severity of their pain on a 100 mm line. The point marked by the patient is measured from the 0 point and the severity of the pain is determined. VAS for children over 7 years old is defined as easy to understand and easy to apply. This scale used in this study will only be evaluated by the child. Studies have shown its validity and reliability. It has been stated that it is suitable for use in all cultures because it is a visual scale.

Wong Baker Faces Pain Comparison Scale (W-BFS) It is one of the most commonly used scales to measure the severity of pain in children. This scale was developed by Donna Lee Wong and Connie Morain Baker in 1981 and revised in 1983. The scale is used in the diagnosis of pain in children aged 3-18 years. It has been reported that the use of W-BPS is safe in children older than three years who can verbally express the degree of pain. There are face shapes and numbers on the scale. Pain is graded between "0" and "10" points. The level of pain felt is expressed with increasing degrees of facial expression. Ask the children "Which face shows your pain?", "How many points would you give your pain?" He will be asked to rate his pain by asking questions such as The parent will also be asked to evaluate the pain according to the child's reaction. Finally, the observer nurse will be asked to rate the pain she observes according to the child's reaction in another environment, without seeing the score given by the child and the parent. It has been stated that it is suitable for use in all cultures because it is a visual scale.

Child Fear Scale (CLO) This scale was developed by McMurtry et al. in 2011. It was translated into Turkish and Turkish validity and reliability study was conducted by Gerceker et al. It is used to measure the level of fear of children. In this method, the child is shown a picture containing five facial expressions evaluated between 0 and 4. 0 indicates no fear; 4 shows the highest fear. These;

* "0 " neutral expression
* "1" very little fear
* "2" some fear (some anxiety)
* "3" more fear (more anxiety)
* "4" is considered the highest possible fear (severe anxiety). This scale can be applied by both the researcher and the family to measure fear before and during the procedure. Before the procedure, children will be told how to use the scale. When the child expresses that he understands, he will be asked to express how afraid he is of the bloodletting. Ask the children, "Can you look at these faces and pick a face that shows how scared you are without blood draw?" You will be asked to score by asking. The score given by the child will be recorded. Likewise, the parent and the observing nurse will be asked to determine the child's fear level without showing it to the child. Finally, after the procedure, the children asked, "Can you choose the face that shows how scared you are during the blood draw?" and will be asked to score according to their facial expressions. The parent will also be asked to rate how scared the child is based on facial expressions, without seeing the child's evaluation during the blood draw. Likewise, the observing nurse will rate the child's fear level and the scores will be recorded. In order to use the scale in this study, the author, who made the Turkish validity and reliability, was contacted via e-mail.

Cognitive-Behavioral Combined Program The Cognitive-Behavioral Combined Program is based on the literature on the subject and taking into account the developmental characteristics of children. Then, opinions were received from experts in the field regarding the program. The program has been updated in line with expert opinions. Five children will be piloted for the implementation of the Cognitive-Behavioral Combined Application Package. The pilot application will be recorded on video and these recordings will be presented to the expert team. Children included in the pilot will not be included in the analysis of the study.

Video Game (Use of Visual and Audio System) In this method, which allows to actively divert attention by giving visual and auditory stimuli together, the focus of attention is drawn to a different place than pain, with the simultaneous activation of many senses. Kaheni et al. (2016) with 80 children with second-degree burns, the children in the experimental group were distracted from pain with a video game during dressing change. It was found that the mean pain score of the children in the experimental group made a significant difference compared to the control group (p<0.05). While 70% of the children in the control group experienced severe pain due to dressing change, most of the children in the experimental group (77.5%) had "some pain".

During the bloodletting process, children in the video game group will be played with audio and visual video games that they can play with one hand. Thus, children will be provided with both visual and auditory stimuli. It will be preferred that children play the video game that they have knowledge about and know how to play the game. For this reason, children in the video game group will be given the chance to choose video games suitable for their age and development level on their parents' smartphones. These video games within the scope of the research will not be named and will not be promoted/advertised.

kaleidoscope Kaleidoscope is a game material in which colorful patterns are seen. When looking inside the kaleidoscope, there are patterns obtained by the reflection of two mirror lights, which are adjacent to each other with an inclination of 60 degrees between them. When the child turns the lower part of the kaleidoscope and looks through the lens, the beads in the kaleidoscope form different patterns. Patterns that appear in different ways attract the child's attention and distract him. In the study of Prajapati (2018), kaleidoscope was found to be effective in reducing pain during blood collection compared to the control group. In the study of Kunjumon and Upendrababu (2018), kaleidoscope was found to be effective in managing pain during intravenous cannulation in children aged 4-6 years. In the research conducted by Semerci and Akgün Kostak (2020), it was determined that the kaleidoscope is effective in reducing pain in children aged 6-12 years. As a result of the research, it was found that distraction cards are more effective in reducing the pain felt than the kaleidoscope.

In this study, a kaleidoscope with colorful patterns that can be used by children with one hand will be used. In the research, the kaleidoscope will be introduced to children and how to use it will be explained. After the procedure, the kaleidoscope will be disinfected using appropriate disinfectant materials.

Data collection will be done on the basis of volunteering to participate in the research. Names of people are not requested and the information obtained from the forms will be kept confidential and will be used only within the scope of this research. Written consent will be obtained for the study and the child and parent will have the right to separate at any stage of the study. The methods to be used in the study do not contain any health risks. When an unexpected situation develops, the studies will be terminated and the necessary intervention will be made.

Ethical and Legal Aspects of Research In order to carry out the research, first of all, permissions were obtained from the authors, who made the Turkish validity and reliability of the scales to be used in the research, via e-mail. The purpose of the study will be explained to the families of the children who meet the research group selection criteria, their questions will be answered and their written consent will be obtained. It will be explained to the parents that the information they give will be kept confidential and will not be used anywhere else. In addition, those who do not want to participate in the study with verbal permission from the children will not be included in the study. In the research, since the use of the human phenomenon requires the protection of individual rights, the relevant ethical principles "Informed Consent Principle", "Volunteering Principle" and "Principle of Protection of Confidentiality" will be fulfilled.

ELIGIBILITY:
Inclusion Criteria:

* Parents and children are willing to participate in the research,
* Written and verbal consent of parents, verbal consent of children,
* The child is in the 8-10 age group,
* The child has come to the center to have blood drawn,
* The child does not have a hearing or auditory problem,
* Absence of pain,
* The child and parent speak and understand Turkish comfortably,
* The child's mental development level to be able to answer the questions asked,
* Not using drugs that will create an analgesic effect in the last 6 hours before the application,
* Children's cognitive level and motor development are suitable for playing video games or using a kaleidoscope,
* Having a video game played by the child on the parent's phone,
* Vascular access is made in one go,
* Vascular access is performed by the same nurse

Exclusion Criteria:

* The child is not in the 8-10 age group,
* The child has a hearing or auditory problem,
* Having pain,
* The child's and parent's inability to speak and understand Turkish comfortably,
* The child is not at the level of mental development to be able to answer the questions asked,
* Parents and children are not willing to participate in the research,
* Parents do not give written and verbal consent, children do not give verbal consent,
* To have used drugs that will create an analgesic effect in the last 6 hours before the application,
* Children's cognitive level and motor development are not suitable for playing video games or using a kaleidoscope,
* Not having a video game played by the child on the parent's phone,
* Vascular access cannot be performed in one go,
* Vascular access is not performed by the same nurse.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Fear average score | 5 minutes
  children' fears before, during and after the procedure will be evaluated (0-4 point).
Pain average score | 5 minutes
  children' pain before, during and after the procedure will be evaluated (0-4 point).
Parents' Satisfaction Level | 5 minutes
  Parents' Satisfaction Level after the procedure will be evaluated (0-4 point).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - KaramanogluMehmetbeyU, Karaman
  - Karamanoglu Mehmetbey University, Karaman

IPD SHARING:
Plan to Share IPD: No